CLINICAL TRIAL: NCT04130633
Title: Behavioral Pharmacology of THC and Alpha-pinene
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: IRB00182689; R01DA043475 (NIH)
Record Dates: First submitted 2019-10-16; First posted 2019-10-17 (Actual); Results first posted 2025-05-22 (Actual); Last update posted 2025-05-22 (Actual); Status verified 2025-05

CONDITIONS: THC; Alpha-pinene
MeSH Terms: interventions — Dronabinol; nabiximols; alpha-pinene

STUDY DESIGN:
Intervention Model Description: All participants will complete all dose conditions (study arms) in a randomized order
Who Masked: Participant, Outcomes Assessor
Masking Description: placebo controlled, double-blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Placebo (Placebo Comparator): Placebo (5mL distilled water)
  Interventions: Drug: Placebo
- Vaporized Pinene (Experimental): 15mg vaporized alpha-pinene
  Interventions: Drug: Alpha-Pinene
- Vaporized THC (Experimental): 30mg vaporized delta-9-THC
  Interventions: Drug: THC
- Vaporized THC and low alpha-pinene (Experimental): 30mg vaporized delta-9-THC and 0.5mg of vaporized alpha-pinene
  Interventions: Drug: THC; Drug: Alpha-Pinene
- Vaporized THC and alpha-pinene (Experimental): 30mg vaporized delta-9-THC and 5mg of vaporized alpha-pinene
  Interventions: Drug: THC; Drug: Alpha-Pinene
- Vaporized THC and high alpha-pinene (Experimental): 30mg vaporized delta-9-THC and 15mg of vaporized alpha-pinene
  Interventions: Drug: THC; Drug: Alpha-Pinene

INTERVENTIONS:
Drug: Placebo — Placebo vapor (distilled water)
  Arms: Placebo
Drug: THC — Pure THC vapor
  Other Names: Cannabis; Delta-9-THC
  Arms: Vaporized THC; Vaporized THC and alpha-pinene; Vaporized THC and high alpha-pinene; Vaporized THC and low alpha-pinene
Drug: Alpha-Pinene — Pure alpha-pinene vapor
  Other Names: Pinene
  Arms: Vaporized Pinene; Vaporized THC and alpha-pinene; Vaporized THC and high alpha-pinene; Vaporized THC and low alpha-pinene

SUMMARY:
This study will evaluate the pharmacokinetics and pharmacodynamics of vaporized alpha-pinene and THC administered via inhalation.

DETAILED DESCRIPTION:
The proposed study will be conducted at the Johns Hopkins Behavioral Pharmacology Research Unit (BPRU). Participants will complete 6 acute drug administration periods in which they will administer THC alone, pinene alone, THC and pinene together, or placebo. Subjective drug effects, cognitive performance, and vital signs will be assessed following drug administration. Each participant will receive all 6 dose conditions in a randomized order using a placebo controlled within-subject crossover design. The study will help the investigators understand the individual and interactive effects of THC and pinene, two common constituents found in cannabis.

ELIGIBILITY:
Inclusion Criteria:

* Have provided written informed consent
* Be between the ages of 18 and 55
* Be in good general health based on a physical examination, medical history, vital signs, 12-lead ECG and screening urine and blood tests
* Test negative for drugs of abuse other than cannabis, including breath alcohol at the screening visit and at clinic admission
* Not be pregnant or nursing (if female). All females must have a negative serum pregnancy test at the screening visit and a negative urine pregnancy test at clinic admission.
* Have a body mass index (BMI) in the range of 18 to 36 kg/m2
* Blood pressure at Screening Visit does not exceed a systolic blood pressure (SBP) of 150 mmHg or a diastolic blood pressure (DBP) of 90 mmHg
* Have no allergies to any of the ingredients used to prepare vapor (THC, pinene).
* Demonstrate competency on cognitive performance measures at screening visit (e.g., PASAT score of 75/90).

Exclusion Criteria:

* Non-medical use of psychoactive drugs other than, nicotine, alcohol, or caffeine 3 month prior to the Screening Visit;
* History of or current evidence of significant medical (e.g. seizure disorder) or psychiatric illness (e.g. psychosis) judged by the investigator to put the participant at greater risk of experiencing an adverse event due to exposure or completion of other study procedures.
* Use of an over-the-counter (OTC), systemic or topical drug(s), herbal supplement(s), or vitamin(s) within 14 days of experimental sessions; which, in the opinion of the investigator or sponsor, will interfere with the study result or the safety of the subject.
* Use of a prescription medication (with the exception of birth control prescriptions) within 14 days of experimental sessions; which, in the opinion of the investigator or sponsor, will interfere with the study result or the safety of the subject.
* Use of dronabinol (Marinol®) within the past month.
* Average use of cannabis more than 2 times per week in the prior 3 months.
* History of clinically significant cardiac arrhythmias or vasospastic disease (e.g., Prinzmetal's angina).
* Abnormal EKG result that in the investigator's opinion is clinically significant.
* Enrolled in another clinical trial or have received any drug as part of a research study within 30 days prior to dosing.
* Having previously sought medical attention to manage adverse effects following acute cannabis use.
* Individuals with anemia or who have donated blood in the prior 30 days

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 33 (Actual)
Dates: Start 2020-11-05 (Actual); Primary Completion 2024-03-08 (Actual); Study Completion 2024-03-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ryan Vandrey, PhD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins University, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Vaporized Delta-9-tetrahydrocannabinol (THC) With and Without Alpha-Pinene: Participants vaporized THC and pinene in a within-subject crossover design:
  1. Placebo
  2. High Pinene (15mg)
  3. High THC (30mg)
  4. High THC (30mg) and Low Pinene (0.5mg)
  5. High THC (30mg) and Mid dose Pinene (5mg)
  6. High THC (30mg and High Pinene (15mg)
Period: Overall Study
Arm/Group | Vaporized Delta-9-tetrahydrocannabinol (THC) With and Without Alpha-Pinene
Started | 33
Placebo | 20
15 mg Alpha-pinene | 22
30mg THC | 20
30mg THC / 0.5mg Pinene | 21
30mg THC / 5mg Pinene | 20
30mg THC / 15mg Pinene | 21
Completed | 19
Not Completed | 14

BASELINE CHARACTERISTICS:
Population: Study completers are reported. 19 participants completed the study.
Groups:
- Vaporized THC With and Without Pinene: All study completers completed the following 6 conditions in a randomized order:
  1. Placebo
  2. High Pinene (15mg)
  3. High THC (30mg)
  4. High THC (30mg) and Low Pinene (0.5mg)
  5. High THC (30mg) and Mid dose Pinene (5mg)
  6. High THC (30mg and High Pinene (15mg)
Arm/Group | Vaporized THC With and Without Pinene
Number analyzed (Participants) | 19
Age, Continuous [Mean (Standard Deviation); unit: years] | 30.57 (8.95)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 11
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 19
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 6
  White | 11
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 19

OUTCOME MEASURES:

1. Primary Outcome: Mean Peak Change From Baseline Drug Effect as Assessed by the Drug Effect Questionnaire (DEQ)
Description: Mean Peak change from baseline rating (0-100) of Drug Effect on the DEQ, a visual analog scale (VAS) self-report questionnaire, with 0 being no effect and 100 being maximum effect.
Time Frame: 0-6 hours, assessed at baseline, 0-hour, and 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 5, and 6 hours post dosing.
Population: Represents study completers
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Vaporized High Alpha-pinene: 15mg of vaporized alpha-pinene
  Alpha-Pinene: Pure alpha-pinene vapor
- Vaporized High THC Alone: 30mg of vaporized pure THC
  THC: Pure THC vapor
- Vaporized High THC and Low Alpha-pinene: 30mg vaporized THC with 0.5mg of vaporized alpha-pinene
  THC: Pure THC vapor
  Alpha-Pinene: Pure alpha-pinene vapor
- Vaporized High THC and Mid-dose Alpha-pinene: 30mg vaporized THC with 5.0mg of vaporized alpha-pinene with
  THC: Pure THC vapor
  Alpha-Pinene: Pure alpha-pinene vapor
- Vaporized High THC and High Alpha-pinene: 30mg of vaporized pure THC and 15mg alpha- pinene
  THC: Pure THC vapor
  Alpha-Pinene: Pure alpha-pinene vapor
Arm/Group | Placebo | Vaporized High Alpha-pinene | Vaporized High THC Alone | Vaporized High THC and Low Alpha-pinene | Vaporized High THC and Mid-dose Alpha-pinene | Vaporized High THC and High Alpha-pinene
Number analyzed (Participants) | 19 | 19 | 19 | 19 | 19 | 19
score on a scale | -1.2 (16.9) | 5.1 (19.7) | 67.2 (27.4) | 66.1 (35.1) | 61.5 (37.0) | 62.9 (38.0)

2. Primary Outcome: Mean Peak Change From Baseline Psychomotor Performance as Assessed by the Digit Symbol Substitution Task (DSST)
Description: Computerized version of Digit Symbol Substitution Task will be administered to assess psychomotor performance. Mean peak change from baseline total correct trials in 90-seconds. Minimum score of 0 but no maximum score (higher scores indicate better performance).
Time Frame: 0-6 hours, assessed at baseline, 0-hour, and 0.5, 1, 1.5, 2, 3, 4, 5, and 6 hours post dosing.
Population: Represents study completers
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | Vaporized High Alpha-pinene | Vaporized High THC Alone | Vaporized High THC and Low Alpha-pinene | Vaporized High THC and Mid-dose Alpha-pinene | Vaporized High THC and High Alpha-pinene
Number analyzed (Participants) | 19 | 19 | 19 | 19 | 19 | 19
score on a scale | 1.6 (10.9) | -4.2 (10.4) | -12.6 (16.9) | -11.2 (13.2) | -8.2 (11.9) | -11.1 (15.8)

3. Primary Outcome: Mean Peak Change From Baseline Working Memory Performance as Assessed by the Paced Auditory Serial Addition Task (PASAT)
Description: Computerized version of Paced Auditory Serial Addition Task administered to assess working memory performance. Mean peak change from baseline total correct trials out of 90 recorded is primary outcome (higher scores indicate better performance).
Time Frame: 0-6 hours, assessed at baseline, 0-hour, and 0.5, 1, 1.5, 2, 3, 4, 5, and 6 hours post dosing.
Population: Represents study completers
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | Vaporized High Alpha-pinene | Vaporized High THC Alone | Vaporized High THC and Low Alpha-pinene | Vaporized High THC and Mid-dose Alpha-pinene | Vaporized High THC and High Alpha-pinene
Number analyzed (Participants) | 19 | 19 | 19 | 19 | 19 | 19
score on a scale | 1.8 (10.3) | 2.5 (12.6) | -8.7 (13.7) | -5.1 (14.7) | -5.7 (11.8) | -7.5 (12.9)

ADVERSE EVENTS:
Time Frame: Up to 6 hours post dose
Description: International Council for Harmonisation (ICH) guidelines are followed for Adverse Event (AE) reporting, as AEs occur they are documented.
Arm/Group | Placebo | Vaporized High Alpha-pinene | Vaporized High THC Alone | Vaporized High THC and Low Alpha-pinene | Vaporized High THC and Mid-dose Alpha-pinene | Vaporized High THC and High Alpha-pinene
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/22 | 0/20 | 0/21 | 0/20 | 0/21
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/22 | 0/20 | 0/21 | 0/20 | 0/21
Other Adverse Events (participants affected / at risk) | 0/20 | 0/22 | 8/20 | 0/21 | 1/20 | 4/21
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=20) | Vaporized High Alpha-pinene (N=22) | Vaporized High THC Alone (N=20) | Vaporized High THC and Low Alpha-pinene (N=21) | Vaporized High THC and Mid-dose Alpha-pinene (N=20) | Vaporized High THC and High Alpha-pinene (N=21)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 2 (2)
Anxiety (Social circumstances) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Tachycardia (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lightheaded (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Fatigue (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-01-18): https://cdn.clinicaltrials.gov/large-docs/33/NCT04130633/Prot_SAP_000.pdf